CLINICAL TRIAL: NCT01230463
Title: Intraoperative Ketorolac Dose of 15 mg Versus the Standard 30 mg on Early Postoperative Pain After Spine Surgery: A Randomised, Blinded, Non-Inferiority Trial
Brief Title: Study of Whether 15 mg Dose of Ketorolac IV is as Effective as a 30 mg Dose.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Kaylene Duttchen, University of Calgary Department of Anesthesia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23237
Record Dates: First submitted 2010-10-27; First posted 2010-10-29 (Estimated); Last update posted 2010-10-29 (Estimated); Status verified 2010-10

CONDITIONS: Pain; Pain, Postoperative
Keywords: Pain, Postoperative; Ketorolac; Anti-Inflammatory Agents, Non-Steroidal; Intraoperative Care
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 15 mg ketorolac IV (Active Comparator)
  Interventions: Drug: Ketorolac Tromethamine
- 30 mg ketorolac IV (Active Comparator)
  Interventions: Drug: Ketorolac Tromethamine

INTERVENTIONS:
Drug: Ketorolac Tromethamine — 15 mg ketorolac IV as a bolus 30 minutes before closure of surgery.
  Other Names: Toradol
  Arms: 15 mg ketorolac IV
Drug: Ketorolac Tromethamine — 30 mg ketorolac IV as a bolus 30 minutes before closure of surgery.
  Other Names: Toradol
  Arms: 30 mg ketorolac IV

SUMMARY:
The primary aim of this study is to show the non-inferiority of 15 mg intraoperative dose of ketorolac as compared to the standard 30 mg ketorolac by looking at the VAS scores 4 hours after an adult spine surgery.

DETAILED DESCRIPTION:
Opioids have traditionally been the cornerstone of acute postoperative pain management. Problematic side effects such as nausea, vomiting, ileus, urinary retention, excess sedation, and respiratory depression are significant disadvantages with the use of opioids. Alternative treatments have been sought. The concept of adding a nonsedating non opioid analgesic agent is appealing and has been validated by previous studies. Nonsteroidal anti-inflammatory drugs (NSAID) are nonsedating and combine analgesic and anti-inflammatory properties ideal for pain after surgery.

Ketorolac is a potent intravenous nonsteroidal anti-inflammatory drug (NSAID), and a non selective cyclooxygenase inhibitor which mediates pain, inflammation and fever. It has been evaluated and used for treatment of moderate to severe pain including postoperative pain. Although intravenous route is not approved by Health Canada, its use is supported in medical literature and clinical practice.

Previous studies have demonstrated the effectiveness of standard 30 mg intravenous ketorolac as an adjunct to opioids for postoperative pain relief. Standard parenteral dose recommended by manufacturer for healthy non elderly population is 30 mg based on a number clinical trials.

Alberta Health Services (AHS) Pharmacy formulary has approved the intravenous use of ketorolac in the dosage range of 10-30 mg depending the patient's weight and medical comorbidities.

NSAIDs, including ketorolac, have an analgesic ceiling effect in which higher doses do not provide any additional pain relief but may increase the likelihood of side effects. Single dose IM ketorolac have been studied in the past showing no difference in analgesia with the 30 and 90 mg dose. Because of risk of drug toxicity and unwanted side effects, patients should be given the lowest effective ketorolac dose. Low dose ketorolac was studied in the adolescents undergoing spine surgery and showed that dose of 0.2mg/kg (11mg) provides supplemental analgesia postoperatively. However, there were no previous studies found on review of the literature using medline search that look at parallel comparison between intraoperative doses of ketorolac in terms of efficacy and safety profile.

ELIGIBILITY:
Inclusion Criteria:

* Patients booked for 1-2 level spine laminectomies and/or decompression
* Adult 18 - 65 years
* Weight of 50 - 110 kg

Exclusion Criteria:

* Previous lumbar laminectomy
* Current anticoagulant use with INR > 1.2
* Narcotic use > 4 weeks
* Known allergy or sensitivity to NSAID or morphine
* Renal insufficiency with creatinine >100 umol/L
* Known liver disease
* History of gastrointestinal bleeding
* Pregnancy, history of bronchial asthma
* NSAID use 2 days before surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Score | Four hours after surgery
  To show the non-inferiority of 15 mg intraoperative dose of ketorolac as compared to the standard 30 mg ketorolac by looking at the VAS scores 4 hours after an adult spine surgery. Minimum clinically significant decrease in VAS pain score is 18 mm.

SECONDARY OUTCOMES:
Morphine Usage After Surgery | 8 hours and 24 hours after surgery
  A 10 mg decrease in morphine use in 24 hours is considered clinically significant.
Morphine Adverse Effects | First 24 hours
  Presence of morphine-related adverse effects such as sedation, nausea, vomiting, respiratory depression, and pruritus.
Postoperative Bleeding | 24 hours after surgery
  Hemoglobin levels will be measured before surgery and 24 hours surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Kaylene Duttchen, MD, Principal Investigator — University of Calgary - Department of Anesthesia; Melinda Davis, MD, Principal Investigator — University of Calgary - Department of Anesthesia
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada